CLINICAL TRIAL: NCT06973564
Title: A Phase 1/2a, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of JAB-23E73 in Adult Patients With Advanced Solid Tumors With KRAS Alteration
Brief Title: JAB-23E73 in Adult Participants With Advanced Solid Tumors With KRAS Alteration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-23E73-1002
Record Dates: First submitted 2025-04-24; First posted 2025-05-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
Keywords: KRAS; KRAS mutation; KRAS G12C, KRAS G12D, KRAS G12V, KRAS G12S, KRAS G12A, KRAS G12D; Pan-KRAS; Targeted Therapy; NSCLC; Pancreas cancer; Colorectal cancer; KRAS-mutant tumor; JAB-23E73
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Phase 1a) (Experimental): Evaluate overall Safety, tolerability, and determine MTD of JAB-23E73 monotherapy.
  Interventions: Drug: JAB-23E73
- Dose Expansion / Optimization Phase (Phase 1b) (Experimental): Determine RP2D of JAB-23E73 in patients with KRAS-alternated NSCLC or other selected tumors
  Interventions: Drug: JAB-23E73
- Indication Expansion (Phase 2a) (Experimental): Evaluate the preliminary antitumor activity of JAB-23E73 monotherapy at the RP2D in patients with advanced or metastatic CRC, PDAC, and other solid tumors.
  Interventions: Drug: JAB-23E73

INTERVENTIONS:
Drug: JAB-23E73 — Oral administration
  Arms: Dose Escalation (Phase 1a)
Drug: JAB-23E73 — Oral administration
  Arms: Dose Expansion / Optimization Phase (Phase 1b)
Drug: JAB-23E73 — Oral administration
  Arms: Indication Expansion (Phase 2a)

SUMMARY:
This study is to evaluate the safety and tolerability of pan-KRAS inhibitor JAB-23E73 in adult participants with advanced solid tumors

DETAILED DESCRIPTION:
Study JAB-23E73-1002 is a multicenter, open-label Phase 1/2a study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anticancer activity of JAB-23E73 as a single agent in adult patients with advanced solid tumors with KRAS alteration. This study consists of a Phase 1a dose-escalation, followed by Phase 1b dose-expansion and Phase 2a indication expansion. After completing dose-escalation, the MTD or preliminary RP2D of JAB-23E73 will be determined. The RP2D will be determined according to the safety, efficacy and PK data from phase 1b. The indication expansion phase will further explore the efficacy and safety in advanced KRAS-alternated tumors which consist of 3 cohorts: Cohort C1, the CRC cohort; Cohort C2, the PDAC cohort; and Cohort C3, other solid tumor cohort.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Participant must be ≥18 years of age at the time of signing the Informed Consent Form (ICF).
* Histologically or cytologically confirmed locally advanced or metastatic solid tumors that are not suitable for curative interventions.
* Patients must have KRAS alterations.
* Participants are required to provide an archived tumor sample.
* Patients with a life expectancy ≥3 months.
* ECOG performance status score of 0 or 1.
* Patients must have at least one measurable lesion as defined by RECIST v1.1.

Exclusion Criteria:

* Inability to swallow oral medications, or presence of gastrointestinal dysfunction or gastrointestinal disorders that may significantly alter the absorption of the study drug.
* Patients who have previously been treated with KRAS G12C inhibitors, KRAS G12D inhibitors, or pan/multi-KRAS inhibitors.
* Known serious allergy to JAB-23E73 or excipient.
* Patients with primary central nervous system tumors.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures or medical intervention.
* QT interval>470 msec.
* LVEF ≤50% assessed by ECHO or MUGA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation (Phase 1a): Determine the Maximum tolerated dose (MTD) of JAB-23E73 monotherapy. | Up to 1 year
  Number and proportion of patients who experience at least 1 dose-limiting toxicity (DLT) during the first 21 days of treatment. A DLT is defined as any toxicities that meet the criteria for a DLT assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 during the evaluation period at any dose.
Dose Escalation (Phase 1a): Evaluate the overall safety and tolerability of JAB-23E73. | Up to 2 years
  Safety and tolerability of repeated cycles from first drug administration up to the Safety Follow Up Visit (SFUV)
Dose Expansion/Optimization (Phase 1b): Determine the Recommended Phase 2 Dose (RP2D) of JAB-23E73 in patients with KRAS- alternated NSCLC or other selected tumors. | Up to 2 years
  RP2D determined by MTD, long term tolerability, PK, efficacy and any other relevant data as available.
Indication Expansion (Phase 2a): Evaluate the preliminary antitumor activity of JAB-23E73 monotherapy at the RP2D in patients with advanced or metastatic CRC, PDAC, and other solid tumors. | Up to 3 years
  ORR, defined as the percentage of patients with the best overall response of confirmed partial response (PR), or complete response (CR) per RECIST v1.1.
Dose Expansion/Optimization (Phase 1b): Determine the RP2D of JAB-23E73 in patients with KRAS- alternated NSCLC or other selected tumors. | Up to 2 years
  RP2D determined by MTD, long term tolerability, PK, efficacy and any other relevant data as available.
Indication Expansion (Phase 2a): Evaluate the preliminary antitumor activity of JAB-23E73 monotherapy at the RP2D in patients with advanced or metastatic CRC, PDAC, and other solid tumors. | Up to 3 years
  ORR, defined as the percentage of patients with the best overall response of confirmed PR, or CR per RECIST v1.1.

SECONDARY OUTCOMES:
Dose Escalation (Phase 1a): Overall Response Rate (ORR) | Up to 2 years
  Objective response rate (ORR) defined as the percentage of patients with the best overall response of confirmed partial response (PR), or complete response (CR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Dose Escalation (Phase 1a): Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) | Up to 2 years
  Cmax of JAB-23E73
Dose Expansion/Optimization (Phase 1b): Overall Response Rate (ORR) | Up to 2 years
  ORR, defined as the percentage of patients with the best overall response of confirmed PR, or CR per RECIST v1.1.
Dose Expansion/Optimization (Phase 1b): Evaluate the overall safety and tolerability of JAB-23E73. | Up to 2 years
  Safety assessments including but not limited to TEAEs, SAEs, deaths and changes in clinical laboratory measures.
Dose Expansion/Optimization (Phase 1b): Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) | Up to 2 years
  Cmax of JAB-23E73

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah